CLINICAL TRIAL: NCT06587308
Title: Effects of Pressure Garments of Varying Designs on Upper Extremity Sensorimotor Functions and Quality of Life After Stroke: A Multicenter, Double-Blind, Prospective Randomized Controlled Trial
Brief Title: Effects of Different Pressure Garments on Upper Extremity Sensorimotor Functions and Quality of Life After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Collaborators: The Affiliated Hospital of Shandong Second Medical University (Unknown); Weifang Municipal People's Hospital (Unknown); Weifang Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JEP-2024-582
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Cerebral Vascular Accident (CVA)/Stroke
Keywords: Pressure Garment; Quality of Life; Stroke Rehabilitation; Occupational Therapy; Motor Activity; Sensory Feedback; Upper Extremity Paresis
MeSH Terms: conditions — Stroke; Motor Activity; Paresis | interventions — S 10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dorsal-Double-Layered 10% Circumferential Reduction (DD-10) Pressure Garment (Experimental): A custom-fabricated finger-to-above-elbow (long glove) pressure garment with 10% of stress. The design is similar to S-10 except it has an extra layer of fabric on the dorsal aspect that gives stronger compression
  Interventions: Other: Dorsal-Double-Layered 10% Circumferential Reduction (DD-10) Pressure Garment
- Single-Layered 10% Circumferential Reduction (S-10) Pressure Garment (Active Comparator): A custom-fabricated single-layered finger-to-above-elbow (long glove) pressure garment with 10% of stress.
  Interventions: Other: Single-Layered 10% Circumferential Reduction (S-10) Pressure Garment
- Single-Layered No Circumferential Reduction (S-0) Pressure Garment (Placebo Comparator): A custom-fabricated single-layered finger-to-above-elbow (long glove) pressure garment with 0% of stress
  Interventions: Other: Single-Layered No Circumferential Reduction (S-0) Pressure Garment

INTERVENTIONS:
Other: Dorsal-Double-Layered 10% Circumferential Reduction (DD-10) Pressure Garment — During Phase IA, i.e., the first four weeks between Time 1 (Baseline) and Time 2 (Week 4), when participants are hospitalized in the rehabilitation department of the hospital. participants will need to wear the DD-10 pressure garment for 3 hours in the morning, 3 hours in the afternoon, and 8 hours at night daily. Additionally, all participants will need to attend an occupational therapy session for 30 minutes, 5 days a week. During Phase IB, i.e., the second four weeks between Time 2 (Week 4), and Time 3 (Week 8), when participants were being discharged from the hospital, they need to continually wearing the pressure garment according to same wearing schedule; however, the participants will not need to attend the occupational therapy session.
  Arms: Dorsal-Double-Layered 10% Circumferential Reduction (DD-10) Pressure Garment
Other: Single-Layered 10% Circumferential Reduction (S-10) Pressure Garment — During Phase IA, i.e., the first four weeks between Time 1 (Baseline) and Time 2 (Week 4), when participants are hospitalized in the rehabilitation department of the hospital. participants will need to wear the S-10 pressure garment for 3 hours in the morning, 3 hours in the afternoon, and 8 hours at night daily. Additionally, all participants will need to attend an occupational therapy session for 30 minutes, 5 days a week. During Phase IB, i.e., the second four weeks between Time 2 (Week 4), and Time 3 (Week 8), when participants were being discharged from the hospital, they need to continually wearing the pressure garment according to same wearing schedule; however, the participants will not need to attend the occupational therapy session.
  Arms: Single-Layered 10% Circumferential Reduction (S-10) Pressure Garment
Other: Single-Layered No Circumferential Reduction (S-0) Pressure Garment — During Phase IA, i.e., the first four weeks between Time 1 (Baseline) and Time 2 (Week 4), when participants are hospitalized in the rehabilitation department of the hospital. participants will need to wear the S-0 pressure garment for 3 hours in the morning, 3 hours in the afternoon, and 8 hours at night daily. Additionally, all participants will need to attend an occupational therapy session for 30 minutes, 5 days a week. During Phase IB, i.e., the second four weeks between Time 2 (Week 4), and Time 3 (Week 8), when participants were being discharged from the hospital, they need to continually wearing the pressure garment according to same wearing schedule; however, the participants will not need to attend the occupational therapy session.
  Arms: Single-Layered No Circumferential Reduction (S-0) Pressure Garment

SUMMARY:
The study aims to compare the effects of dorsal-double-layered 10% circumferential reduction (DD-10), single-layered 10% circumferential reduction (S-10), and single-layered no circumferential reduction (S-0) pressure garments on sensorimotor functions, including motor control, dexterity, muscle tone, pain, self-perceived upper extremity function, and quality of life among stroke patients during the 8 weeks of application (Time 1: Baseline, Time 2: Week 4, Time 3: Week 8).

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 80 years of age
* Within 1-12 months of ischemic or hemorrhagic stroke
* First onset resulting in hemiparesis of a limb with Burnnstrom stage of 3, 4 or 5
* Modified Ashworth Scale with scores of less than or equal 2 for elbow, wrist, and hand muscle tone in the affected upper extremity
* Able to understand instruction

Exclusion Criteria:

* Serious cardiovascular or respiratory diseases
* Skin lesions, infections or other skin problems
* Serious circulatory problems such as deep vein thrombosis
* Allergies or significant discomfort to pressure garment materials
* Upper extremity fractures or severe joint problems
* Severe cognitive impairment with Saint Louis University Mental Status (SLUMs) scores equal to or less than 27 (above high school level of education)/25 (below high school level of education)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) | Baseline, Week 4. Week 8
  A classic tool used to assess the rehabilitation process of stroke patients from the aspects of sensorimotor function and level of life activities. It has two main domains, i.e., upper extremity and lower extremity. The 33-item upper extremity domain that will be used in this study includes the range of motion of the shoulder, elbow, wrist, and fingers as well as elements such as grip strength and hand coordination. Scored between 0 and 66, higher scores indicating greater function.

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | Baseline, Week 4. Week 8
  A method used to assess muscle tone or muscle spasticity. It uses a scale of 0 to 4, where 0 indicates no spasticity and 4 indicates severe spasticity.
Visual Analogue Scale (VAS) | Baseline, Week 4. Week 8
  A 10-cm pain scale with one end of the scale represents no pain and the other end represents unbearable pain. Subjective perception of pain is obtained by drawing a vertical line between these two endpoints.
Box and Block Test (BBT) | Baseline, Week 4. Week 8
  A quantitative tool used to assess upper extremity sensorimotor function, including hand coordination, dexterity, speed of movement, and fine hand movements. Assessment is done by transferring a set of cubes from one side of a box separated into two equal-sized compartments (by a divider) to the other side within one minute.
Disabilities of Arm, Shoulder and Hand (DASH) Outcome Measure | Baseline, Week 4. Week 8
  A widely used tool for assessing upper extremity function. Its disability/symptom module has 30 items that covers a wide range of functional daily activities. Scored between 0 and 100, higher scores indicating more severe disability.
36-Item Short Form Health Survey (SF-36) | Baseline, Week 4. Week 8
  A 36-item survey questionnaire designed to provide insight into health status and quality of life of an individual, allowing comprehensive assessment of physical, psychological, and social functioning. Each dimension is converted into a score of 100 points by assigning weights to the entries according to the degree to which they affect the quality of life. The level of the score directly reflects the health status, with higher scores indicating better functional status and quality of life in this area.

OTHER OUTCOMES:
Brunnstrom Recovery Stage (BRS) | Prior to participant enrolment
  A brief and easy-to-administer measure used to assess motor function. It consists of three items for the arm (BRS-A), hand (BRS-H), and leg (BRS-L), all of which are scored on a 6-point Likert-type scale, with each stage representing a different motor characteristic and change in muscle control.
Modified Ashworth Score (MAS) | Prior to participant enrolment
  A method used to assess muscle tone or muscle spasticity. It uses a scale of 0 to 4, where 0 indicates no spasticity and 4 indicates severe spasticity..
Saint Louis University Mental Status (SLUMS) Examination | Prior to participant enrolment
  A measure used to assess cognitive functioning. It assesses several cognitive domains such as attention, memory, executive functioning, orientation, and numeracy. Specific items include vocabulary learning, memory recall, numeracy, clock drawing, number reversal, and image naming. It is scored on a 30-point scale, with higher scores indicating better cognitive functioning and lower scores suggesting impaired cognitive functioning. Items are designed to cover multiple cognitive domains to provide a more comprehensive assessment.

CONTACTS AND LOCATIONS:
Overall Officials: SIaw Chui Chai, PhD, Principal Investigator — Occupational Therapy Programme, Centre for Rehabilitation and Special Needs Studies (iCaRehab)
Locations (3):
- China (3):
  - The Affiliated Hospital of Shandong Second Medical University, Weifang, Shandong
  - Weifang Hospital of Traditional Chinese Medicine, Weifang, Shandong
  - Weifang Municipal Peoples Hospital, Weifang, Shandong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu Z, Chai SC, Chu SY, Li K. Effects of pressure garments of varying designs on upper extremity sensorimotor functions and quality of life after stroke: Study protocol for a multicenter, double-blind, prospective randomized controlled trial. PLoS One. 2025 Jun 23;20(6):e0326680. doi: 10.1371/journal.pone.0326680. eCollection 2025. PMID 40549786